CLINICAL TRIAL: NCT05812235
Title: Bone Microstructure by Using High-resolution Peripheral Quantitative Computed Tomography After Esophagectomy
Brief Title: Bone Microstructure by Using HR-pQCT After Esophagectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Nagasaki University (Other)
Responsible Party: Principal Investigator, Kobayashi Shinichiro, Surgery, Nagasaki University
Other Study IDs: NagasakiU3
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Osteoporosis; Sarcopenia; Esophageal Cancer
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Protein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Esophagectomy: 48 patients with esophagectomy due to esophageal cancer before no more than 3 years
  Interventions: Procedure: esophagectomy
- Healthy Control: 70 patients without gastrectomy , who are similar background in other group, are collected from date Pathologic analysis of primary osteoporosis: investigating age and osteoporosis related changes of bone microstructure by using HR-pQCT (UMIN000023535)

INTERVENTIONS:
Procedure: esophagectomy — esophagectomy
  Groups: Esophagectomy

SUMMARY:
Esophagectomy is most curative treatment to esophageal cancer. However, osteoporosis , which is characterized by both the loss of bone mass and the deterioration of bone architecture, is a serious complication in the long course after surgery. The aim of the present study was to evaluate osteoporosis by using high-resolution peripheral quantitative computed tomography (HR-pQCT) in the long course after esophagectomy. At least 3 years should have elapsed since operation without recurrence of esophageal cancer.

DETAILED DESCRIPTION:
The patients after esophagectomy loss appetite and decrease the weight. Esophagectomy especially cause severe sarcopenia and metabolic change. Osteoporosis, which is characterized by both the loss of bone mass and the deterioration of bone architecture, is a serious complication in the long course after esophagectomy. The primary tools for assessing volumetric density and bone structure are quantitative computed tomography (QCT) and more recently, high-resolution peripheral quantitative computed tomography (HR-pQCT). However the validation of osteoporosis with HR-pQCT in the long course after esophagectomy remain elusive. The aim of the present study was to evaluate osteoporosis by using HR-pQCT in the long course after esophagectomy. At least 3 years should have elapsed since esophagectomy without any recurrence.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 years have elapsed since esophagectomy due to esophageal cancer
* Provide signed informed consent

Exclusion Criteria:

* Current use of the following osteoporosis agents; Teriparatide, Denosumab, and - -
* bisphosphonate
* Present malignancy (except in situ carcinoma)
* Radiotherapy
* Any condition that required chronic (greater than three months cumulative and greater than 5 mg/day) glucocorticoid therapy
* Other diseases which affect bone metabolism Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures Received > 3 months (or equivalent) of osteoporosis treatment Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Japanese
Sampling Method: Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparing bone microstructure in control and Esophagectomy groups | 1day
  volumetric bone mineral density

SECONDARY OUTCOMES:
Comparing bone microstructure with serum biomarkers of osteoporosis | 1day
  Correlation between bone mineral density in esophagectomy and biomarkers (25-hydroxyvitaminD, calcium, iPTH, P1NP, ICTP, TRACP5b)
Comparing bone microstructure with dual-energy X-ray absorptiometry | 1day
  Correlation of bone mineral density between esophagectomy and DXA

IPD SHARING:
Plan to Share IPD: No